CLINICAL TRIAL: NCT00458172
Title: Study 1 of Lay Theories of Health: Conceptualizations of Physical, Mental, and Social Health in Young and Middle-Aged Adults
Brief Title: Lay Theories of Health in Young and Middle Aged American Adults
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: Blue Cross Blue Shield of Michigan Foundation (Other)
Responsible Party: Principal Investigator, Christina A. Downey, Ph.D. Student, University of Michigan
Other Study IDs: HUM00011805
Record Dates: First submitted 2007-04-04; First posted 2007-04-09 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Healthy
Keywords: lay theories; health concepts; survey; internet research; Ideas about health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Assessment of beliefs and attitudes

SUMMARY:
This study is the second empirical investigation in a series of studies, examining what everyday people believe that it means to be healthy. Part of this research also involves examining whether these lay theories of health vary according to various demographic classifications.

DETAILED DESCRIPTION:
In the journal "Science," Engel (1977) proposed the term "biopsychosocial model" to recognize the social and psychological factors impacting health and illness. Psychologists have played a significant role in contributing to current evidence for this model, including understanding how individuals think about their health.

Work in this area has corresponded to work on the implicit theories of individuals, and how those implicit theories have an impact upon cognition, affect, and behavior. Implicit theories are mental constructions about specific phenomena which, while often elaborate in structure, content, and function, are not well articulated by those who hold them.

A failure to thoroughly investigate lay theories of health has implications for the biopsychosocial model of health and illness, which states that it is not only the knowledge of the physician, but also the beliefs of the patient, that have consequences for the patient's experience of health and illness. Research on individual beliefs regarding illness has been accumulating for some time, and it is becoming apparent that these beliefs have significant consequences for individual health behavior. However, current studies assessing lay theories regarding illness may be inadequate to achieving the goal of fully learning how lay theories have an impact upon health. The methodologies utilized rarely distinguish whether the implicit theories under study should be attributed to laypeople or to experts, and tend to assume that health and illness have perfect reciprocal correspondence with one another in the minds of laypeople. If researchers hope to understand laypeople's theories about health, exclusively investigating lay theories of illness will not suffice to answer the question.

The present series of studies seeks to investigate a number of unanswered questions in the existing literature on lay theories of health. In a Prestudy, we investigated how adult laypeople define what it is to be healthy through open-ended survey questions. At the present time (the focus of the current IRB application) we hope to have participants rate the importance of each of the previously-gathered items to their concept of health (Study 1). We will then present the most important items in pairs to a second sample, and ask those participants to rate how similar or dissimilar the items are to one another. From these ratings, we will determine the structure of lay theories of health through scaling procedures. After determining the structure of lay theories (e.g., in terms of dimensions), we will focus on developing a comprehensive measure of lay theories of health. We will at that time conduct a series of validation studies to determine whether and how these dimensions of lay theories differ from those of experts, do or do not correspond with existing constructs measuring well-being, and are utilized by laypeople in making health judgments and decisions (which will be reviewed and conducted at a later date).

ELIGIBILITY:
Inclusion Criteria:

* English primary language
* U.S. residency (but not necessarily citizenship)

Exclusion Criteria:

* Only by age

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 302 (Actual)
Dates: Start 2007-04; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina A Downey, M.S., Principal Investigator — University of Michigan
Locations (1):
- Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study website - please click link to participate in this 15-minute study now. — https://www.psychdata.com/s.asp?SID=121042